CLINICAL TRIAL: NCT03768869
Title: Fever and Neutropenia in Pediatric Oncology Patients: A Randomized, Controlled, Multi-Center Study of Outpatient Therapy Evaluation of Genomic and Proteomic Correlates
Brief Title: Fever and Neutropenia in Pediatric Oncology Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient data to answer the study question
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 05-0300.cc
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Fever; Neutropenia
Keywords: Pediatrics; Oncology; Outpatient therapy
MeSH Terms: conditions — Fever; Neutropenia; Neoplasms | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Patients will be stratified as high risk, where they will receive inpatient management, or low risk, where they will then be randomize to receive inpatient or outpatient management.
Masking Description: Because inpatient management and outpatient management use different treatment methods, blinding is not possible.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Risk: Oupatient Management (Experimental): Patients will be categorized according to risk of serious bacterial infection per risk stratification system, which is based on demographic, clinical history and physical findings that have been shown to be predictive of risk.
  Interventions: Drug: Low Risk: Oupatient Management
- Low Risk: Inpatient Management (Active Comparator): Patients will be categorized according to risk of serious bacterial infection per risk stratification system, which is based on demographic, clinical history and physical findings that have been shown to be predictive of risk.
  Interventions: Drug: Low Risk: Inpatient Management
- High Risk: Inpatient Management (Active Comparator): Patients will be categorized according to risk of serious bacterial infection per risk stratification system, which is based on demographic, clinical history and physical findings that have been shown to be predictive of risk.
  Interventions: Drug: High Risk: Inpatient Management

INTERVENTIONS:
Drug: Low Risk: Oupatient Management — Intravenous Levaquin initially, then oral dosing. Patient discharged to go home to finish medication cycle after initial 120 minutes observation. Patients will be evaluated daily in the clinic, and his or her temperature must be taken and recorded four times per day. Blood cultures will be drawn at clinic visits.
  Other Names: Oral Antibiotics
  Arms: Low Risk: Oupatient Management
Drug: Low Risk: Inpatient Management — Broad spectrum intravenous antibiotics. Daily blood work will be drawn, and patients will be monitored for fever and neutropenia in hospital.
  Other Names: IV Antibiotics
  Arms: Low Risk: Inpatient Management
Drug: High Risk: Inpatient Management — Broad spectrum intravenous antibiotics. Daily blood work will be drawn, and patients will be monitored for fever and neutropenia in hospital.
  Other Names: IV Antibiotics, High Risk
  Arms: High Risk: Inpatient Management

SUMMARY:
It is possible to distinguish between pediatric oncology patients who are at high or low risk for serious infection during periods of fever and treatment related neutropenia based on clinical parameters. Patients with low risk can be safely treated as outpatients primarily using oral antibiotics. It is possible to improve methods of risk stratification through the addition of genomic and proteomic factors.

DETAILED DESCRIPTION:
Outpatient management of patients considered to be at low risk for serious bacterial infection has been explored using risk stratification schema based on clinical parameters. First, patients will be stratified based on a clinical risk stratification schema. Patients stratified to the low risk group will be randomized between treatment using standard inpatient intravenous antibiotic therapy or outpatient antibiotic therapy using primarily an oral regimen. Second, an evaluation of proteins important to the innate immune system will be performed to provide a molecular characterization of episodes based on etiology. Third, single nucleotide polymorphisms in genes important for innate immunity will be evaluated to determine effect of each on infection risk during treatment induced neutropenia. Finally, we will develop a bank of both plasma and DNA specimens correlated with clinical outcomes for future use.

ELIGIBILITY:
Inclusion Criteria:

1. Any pediatric patient age <21 years with an oncology diagnosis who is undergoing therapy and is expected to have treatment related neutropenia.

Exclusion Criteria:

1. Any patient who has previously undergone autologous or allogeneic bone marrow transplant will be excluded from study enrollment. If a patient is expected to undergo autologous or allogeneic bone marrow transplant as part of therapy at some point after enrollment in the study he/she will be removed from the study at the start of their bone marrow transplant.
2. Any patient with a documented allergy to Levofloxacin or any other fluoroquinolone will be excluded.
3. Patients with a known pregnancy will be excluded.
4. Any patient with an underlying chronic musculoskeletal condition (ie Juvenile rheumatoid arthritis, Systemic lupus erythematosis etc) which may make evaluation for joint toxicity related to quinolone treatment difficult.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2009-04-03 (Actual); Study Completion 2009-04-03 (Actual)

PRIMARY OUTCOMES:
Low Risk Treatment | Start of study to end of study, up to two years
  The response to initial antibiotic management without modification with regards to resolution of the episode of fever and neutropenia, measured through blood cultures
Protein Evaluation | Start of study to end of study, up to two years
  Comparison of the level of each protein at the initiation of each episode versus resolution to determine if there is a pattern of proteins that correlates with an infectious outcome, measured using ELISA techniques
Genomics Evaluation | Start of study to end of study, up to two years
  A comparison of proven infections between patients with the wild-type and variant forms of each gene studied, taken through DNA specimens

SECONDARY OUTCOMES:
Cost Benefit Analysis | Start of study to end of study, up to two years
  A cost-benefit analysis between the arms, duration of fever per episode between the arms, and number of admissions or deaths. Medical cost will be obtained through billing records and indirect costs will be estimated through information obtained from the family.
Protein Evaluation | Start of study to end of study, up to two years
  Determine trends of protein markers on days 3 and 5 of evaluation, using ELISA techniques.
Genomics Evaluation | Start of study to end of study, up to two years
  A comparison of the number of episodes of fever and neutropenia per patient and the duration of fever per episode between the wild type and variant forms of each gene, taken through DNA specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Maloney, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States